CLINICAL TRIAL: NCT03294239
Title: Transurethral Versus Percutaneous Endoscopic Management of Bladder Stones in Boys: A Comparative Prospective Randomized Study
Brief Title: Transurethral Versus Percutaneous Endoscopic Management of Bladder Stones in Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Alaa, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUEMBS
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-09

CONDITIONS: Pediatric Bladder Stones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Transurethal group) (Experimental): Patients will have trans urethral approach for management of their bladder stones. Either pneumatic or Holmium:YAG laser will be used for stone disintegration. Stone basket and/or Elics current evacuation will be used to retrieve stone fragments. Urethral catheter will be applied for 48 hours.
  Interventions: Procedure: Transurethral extraction of bladder stone(s)
- Group B (Percutaneous group) (Experimental): Patients will have per cutaneous approach for management of their bladder stones. After initial cystoscopy a Foley's urethral catheter will be fixed for continuous irrigation. Then, the bladder will be filled to capacity with normal saline. Access to the distended bladder will be obtained by 10-gauge needle in the mid line 1-2 cm above the pubic bone. Once suitable placement is confirmed with return of fluid, a guide wire will be passed through the needle into the bladder. Dilatation will be done using 8-10 Fr coaxial dilators then single fascial dilator with placement of 16 Fr Amplatz sheath as a working tract. No ultrasonic or fluoroscopic guidance will be used. Stone basket will be used to extract the stone. If the stones were larger than the used sheath, disintegration will be performed with a pneumatic lithotrite. Primary skin closure of the suprapubic stab wound by one stitch will be done and the urethral catheter will remain for 48 hours.
  Interventions: Procedure: percutaneous extraction of bladder stone(s)

INTERVENTIONS:
Procedure: Transurethral extraction of bladder stone(s) — Patients will have transurethral approach for management of their bladder stones. Either pneumatic or Holmium:YAG laser will be used for stone distentegration. Stone basket and/or Elics current evacuation will be used to retrieve stone fragments. Urethral catheter will be applied for 48 hours.
  Arms: Group A (Transurethal group)
Procedure: percutaneous extraction of bladder stone(s) — Patients will have percutaneous approach for management of their bladder stones. After initial cystoscopy a Foley's urethral catheter will be fixed for continuous irrigation. Then, the bladder will be filled to capacity with normal saline. Access to the distended bladder will be obtained by 10-gauge needle in the midline 1-2 cm above the pubic bone. Once suitable placement is confirmed with return of fluid, a guide wire will be passed through the needle into the bladder. Dilatation will be done using 8-10 Fr coaxial dilators then single fascial dilator with placement of 16 Fr Amplatz sheath as a working tract. No ultrasonic or fluoroscopic guidance will be used. Stone basket will be used to extract the stone. If the stones were larger than the used sheath, disintegration will be performed with a pneumatic lithotrite. Primary skin closure of the suprapubic stab wound by one stitch will be done and the urethral catheter will remain for 48 hours.
  Arms: Group B (Percutaneous group)

SUMMARY:
To compare safety and efficacy of trans urethral and per cutaneous approaches in endoscopic management of bladder stones in boys younger than 14 years

DETAILED DESCRIPTION:
Pediatric urolithiasis remains endemic in developing nations, affecting children at ages less than 1 year to adolescence. The prevalence rate is high at 5% to 15% compared with 1% to 5% in developed countries. Recent studies have shown that the percentage of bladder stones in pediatric urolithiasis is 30%.

Open cystolithotomy has been the traditional modality to treat bladder stones. It has the inherent problems of a long scar, prolonged catheterization and hospitalization and risk of wound infection .The advent of improved endoscopic techniques in the form of gradual decrease in endoscopic sizes and the development of effective lithotripters have made trans urethral endoscopic management of bladder stones feasible. Excellent stone-free rates with trans urethral lithotripsy with minimal complications make it a preferred treatment option . However, in children especially boys, the small caliber of urethra raise concerns about the ability of stone fragments clearance and the possibility of iatrogenic urethral stricture occurrence. This renders trans urethral cystolithotripsy to be more difficult and unfavorable .

Per cutaneous cystolithotomy (PCCL) can be a safe alternative with low morbidity and complication rate. It has been performed safely for bladder stones up to 5 cm in size. This procedure may carry many advantages in the form of short operative time, more feasible stone fragments retrieval and less need for stone disintegration with its possible sequel as mucosal perforation or stone escaping inside the bladder that prolong the operative time.

On the other hand PCCL has important disadvantages such as the presence of an incision, the need to dilate a tract and the potential need for a urethral catheter or supra pubic tube. There are other reported complications including paralytic ileus, abdominal distention from escape of irrigating fluid into the abdominal cavity and urine leakage. It also carries a risk of bowel injury especially if there is a history of abdominal or pelvic surgery.

To the best of our knowledge, no previous prospective studies compared between per cutaneous and trans urethral approaches for endoscopic management of bladder stones in male children.

The aim of the study is to compare safety and efficacy of trans urethral and per cutaneous approaches in endoscopic management of bladder stones in boys younger than 14 years.

ELIGIBILITY:
Inclusion Criteria:

* Boys less than 14 yrs old age with bladder or urethral stones less than 3 cm.

Exclusion Criteria:

* Neurogenic bladder. Augmented bladder. Upper urinary tract stones that needs simultaneous ureteroscopy, PNL or ureteral stent insertion.

Bleeding tendency. Urethral stricture. Stone in fossa navicularis that can be extracted after meatotomy.

Ages: 1 Month to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
stone free state | 1 week post operative
  The number of patients with no residual stone fragments with no need to shift to other modality or auxiliary maneuver

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided